CLINICAL TRIAL: NCT00001065
Title: A Phase II Trial of Amphotericin B Oral Suspension for Fluconazole-Resistant Oral Candidiasis in HIV-Infected Patients
Brief Title: A Study of Amphotericin B in the Treatment of Fungal Infections of the Mouth in HIV-Infected Patients Who Have Not Had Success With Fluconazole
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 295; 11271 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Candidiasis, Oral; HIV Infections
Keywords: Administration, Oral; Acquired Immunodeficiency Syndrome; Amphotericin B; AIDS-Related Complex; Candidiasis, Oral; Suspensions
MeSH Terms: conditions — Candidiasis, Oral; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Amphotericin B

INTERVENTIONS:
Drug: Amphotericin B

SUMMARY:
To assess response and toxicity in patients with fluconazole-resistant oral candidiasis ( thrush ) when given initial induction with amphotericin B oral suspension.

Experience with amphotericin B oral suspension for drug-sensitive thrush in HIV-infected patients is limited but encouraging.

DETAILED DESCRIPTION:
Experience with amphotericin B oral suspension for drug-sensitive thrush in HIV-infected patients is limited but encouraging.

Patients swish and swallow amphotericin B oral suspension after each meal and at bedtime for 14 days, at which time they are deemed a responder, nonresponder, or failure to induction therapy. Responders receive maintenance twice daily, while nonresponders receive 14 further days of initial induction. Failures discontinue the study. Responders after 28 days of induction are placed on maintenance. After successful completion of initial induction, patients remain on study for 6 months.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection OR diagnosis of AIDS.
* Diffuse oral candidiasis, symptomatic or asymptomatic, that is resistant to fluconazole.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Current symptoms of esophageal candidiasis unless there are negative endoscopic visualization and biopsy for Candida or related yeasts.
* Perioral lesions only (e.g., angular stomatitis, perleche).
* Inability to swish and swallow oral solution.
* Inability to tolerate further oral therapy for thrush.

Concurrent Medication:

Excluded:

* Fluconazole.
* Itraconazole.
* Ketoconazole.
* Flucytosine.
* Intravenous amphotericin or other non-study formulations.
* Nystatin.
* Clotrimazole.
* Other investigational antifungal agents.
* Systemic cytotoxic chemotherapy for malignancy.

Concurrent Treatment:

Excluded:

* Radiation therapy to the mouth, neck, or chest.

Patients with the following prior conditions are excluded:

* Esophageal candidiasis, proven or presumptive, occurring since fluconazole failure.
* Successful treatment of thrush with fluconazole at <= 200 mg/day after original treatment failure.
* History of oral candidiasis that recurred or persisted despite IV amphotericin B given once or more weekly.
* History of anaphylaxis to amphotericin B.
* History of hypersensitivity to components in amphotericin B oral suspension.

Prior Medication:

Excluded within 6 weeks prior to study entry:

* Cytotoxic therapy for malignancy.
* Corticosteroids at higher than replacement doses.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70
Dates: Study Completion 1998-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zingman BS, Study Chair; Wheat LJ, Study Chair
Locations (32):
- United States (30):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Howard University Hosp., Div. of Infectious Diseases, ACTU, Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS, Miami, Florida
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Weiss Memorial Hosp., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico
- Mbeya Med. Research Program, Mbeya Referral Hosp. CRS, Mbeya, Tanzania